CLINICAL TRIAL: NCT01368952
Title: Efficacy Study of Pure Prone Positioning Therapy in Patients With Mild to Moderate Obstructive Sleep Apnea
Brief Title: The Effect of Pure Prone Positioning Therapy for the Patients With Mild to Moderate Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Arman Afrashi, MD., Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IGHCEAH-IRB-286; 286 (Other: IRB Number of IGHCEAH)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Prone positioning; Positional Treatment; Hypoxemia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pure Prone Positioning (Active Comparator): Sleeping in prone position by pure prone positioning device, which consisted of a pillow mounted on a table designed to keep the subjects sleeping prone.
  Interventions: Device: Pure prone positioning
- Baseline (No Intervention): No intervention for sleep position

INTERVENTIONS:
Device: Pure prone positioning — Pure prone positioning device consisted of a pillow mounted on a table designed to keep the subjects sleeping prone.
  Other Names: Positional treatment
  Arms: Pure Prone Positioning

SUMMARY:
Efficacy of Pure Prone Positioning (PPP) treatment in improving apnea-hypopnea index (AHI) and nocturnal oxygen saturation was investigated in mild to moderate Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
Sleeping in prone position could be effective in the management of obstructive sleep apnea (OSA) by reducing the gravity effect on the upper airway and hence collapsibility. Pure prone positioning (PPP) consisted of a pillow mounted on a table designed to keep the subjects sleeping prone with the head extended in line with the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled to the study among one hundred and eighty-four consecutive patients who were admitted to our sleep center with 6 beds in a tertiary care hospital, during 3 months period. Of these, 36 patients with mild to moderate OSA (AHI=5-30 events/h) were invited to participate in the study based on the selection criteria, and 29 patients with mild to moderate OSA on their baseline PSG, (17 males, 12 females) gave informed consent and participated in the study.

Exclusion Criteria:

* Patients having BMI>35 and/or abdominal and/or trunkal obesity that may hinder prone sleeping , upper airway pathology (nasal polyp, nasal turbinate hypertrophy, chronic sinusitis, nasal septum deviation, upper airway infection, Mallampati score and tonsil size grade of IV), any other concomitant sleep disorder (narcolepsy, periodic leg movement syndrome, insomnia, sleep related hypoventilation-hypoxemia and central sleep apnea syndrome), psychiatric disorder such as panic disorder, heart failure and coronary artery disease were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | ''Baseline PSG night'' and ''pure prone positioning night within two weeks of baseline PSG night''
  Reduction in AHI during pure positioning night as compared to baseline night

SECONDARY OUTCOMES:
Nocturnal oxygen saturation | ''Baseline PSG night'' and ''pure prone positioning night within two weeks of baseline PSG night''
  Comparison of mean oxygen saturation, minimum oxygen saturation and proportion of time spent during sleep with oxygen saturation below 90% (as measures of nocturnal hypoxemia) in pure prone positioning night with that of the baseline night.
Sleep efficiency | ''Baseline PSG night'' and ''pure prone positioning night within two weeks of baseline PSG night''
  Improvement in sleep efficiency in prone positioning night as compared to baseline night.

CONTACTS AND LOCATIONS:
Overall Officials: Arman Afrashi, MD, Principal Investigator — The Department of Otolaryngology-Head and Neck Surgery, Izmir Dr Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Turkey; Zeynep Z Ucar, MD, Study Director — The Department of Sleep Disorders, Izmir Dr Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Turkey
Locations (1):
- The Department of Sleep Disorders, Izmir Dr Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] George CF, Millar TW, Kryger MH. Sleep apnea and body position during sleep. Sleep. 1988 Feb;11(1):90-9. doi: 10.1093/sleep/11.1.90. PMID 3363274
- [Result] Matsuzawa Y, Hayashi S, Yamaguchi S, Yoshikawa S, Okada K, Fujimoto K, Sekiguchi M. Effect of prone position on apnea severity in obstructive sleep apnea. Intern Med. 1995 Dec;34(12):1190-3. doi: 10.2169/internalmedicine.34.1190. PMID 8929648